CLINICAL TRIAL: NCT02873793
Title: Analysis of Transposon Control Pathways in Germinal Cancers of the Testicle
Acronym: SEMINOMES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: FAUQUE 2014
Record Dates: First submitted 2016-08-04; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-07

CONDITIONS: Germinal Cancers of the Testicle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Extraction of total RNA from healthy and tumour tissues

GROUPS / COHORTS (3):
- 7/8 cases pure seminomas
  Interventions: Genetic: Extraction of total RNA from healthy and tumour tissues
- 5 cases of non-seminoma
  Interventions: Genetic: Extraction of total RNA from healthy and tumour tissues
- 3 cases of composite tumours seminoma/non-seminoma.
  Interventions: Genetic: Extraction of total RNA from healthy and tumour tissues

INTERVENTIONS:
Genetic: Extraction of total RNA from healthy and tumour tissues

SUMMARY:
By analogy with the mouse, the activity of control pathways for transposable elements (TE) in foetal primordial germinal cells could prove to be a determinant for fertility in adulthood in humans. Moreover, defects in the control of transposable elements (TE) could also contribute to the aetiology of germinal testicular cancer, by inducing chromosomal instability and tumorigenesis. In this context, the aim is to analyse a specific type of adult germinal testicular cancers, seminomas. Directly related to our research interest, the histological, transcriptomic and epigenetic features of theses adult tumours are reminiscent of germinal cells normally present in foetuses. The investigator postulates that these similarities could also extend to the biology of transposable elements (TE), and in particular to the initiation of the control of these elements. The management of seminomas requires surgery, orchiectomy, which consists of the total excision of the affected testicles. Using high-resolution high-throughput sequencing techniques, we propose to analyse the control pathways of transposable elements (TE) in tumour samples harvested from surgical pieces in comparison with adjacent healthy tissue. The results obtained in these tumour samples will be compared with those in normal foetal gonad samples.

ELIGIBILITY:
Inclusion Criteria:

* men who have provided oral consent
* men with germinal testicular cancer with negative or low serum markers (Alpha Foeto Protein AFP and Human Chorionic Gonadotrophin hCG), indicators of a seminomatous-type tumour
* men who have undergone orchiectomy (total excision of the affected testicle)
* confirmation of the diagnosis of seminomatous or non-seminomatous type by histology of the surgical piece
* absence of hepatitis B or C or infection with human immunodeficiency virus (HIV).

Exclusion Criteria:

* men without national health insurance cover
* Adults under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men with germinal testicular cancer
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
The role of Transposable Element in tumorigenesis seminomas adults | through the study completion up to 36 months
  Transcriptomic analysis of adult seminomas

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France